CLINICAL TRIAL: NCT03400748
Title: ANET Electrosurgery Applicator Pilot Evaluation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: business reason
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 15
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Results first posted 2021-09-27 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer; Lung Cancer Metastatic
Keywords: Electrosurgery; RF ablation; Minimally invasive; Lung cancer; Lung metastasis; Lung tumor; Primary; Metastatic; Endobronchial ultrasound; EBUS
MeSH Terms: conditions — Lung Neoplasms; Hyperthermia; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- RF Ablation (Experimental): Single-arm study where subjects receive RF ablation prior to a scheduled surgical resection.
  Interventions: Device: RF Ablation

INTERVENTIONS:
Device: RF Ablation — The intervention consists of a bronchoscopic approach to ablate lung tumors with radio-frequency energy.

SUMMARY:
Evaluate the preliminary safety and performance of the Electrosurgery Applicator (ANET device) during and after bronchoscopic ablation of a target pulmonary nodule/tumor.

DETAILED DESCRIPTION:
This study is a prospective, single arm, single center study that will evaluate the effectiveness of the ANET Electrosurgery Applicator in up to 10 subjects.

Subjects who consent to participate in this study will have a lung tumor that is scheduled to be removed surgically as part of their normal treatment. During the surgical procedure, just prior to resection the subject's tumor will be treated with the ANET device. The ANET device uses a bronchoscope to reach the tumor. Ultrasound on the bronchoscope, CT, and X-rays are used to make sure the ANET device is in the tumor. Once in the tumor, the ANET device uses radio-frequency (RF) ablation to treat the tumor. After standard surgical resection the tumor and surrounding tissue is evaluated to characterize the effect of the ANET.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with Stage I or Stage II primary lung cancer or metastatic lung tumor
2. Pathological proof of target nodule/tumor type and malignancy
3. Target nodule/tumor which can be accessed via EBUS bronchoscopy
4. Resection/surgical candidate
5. Participants must be at least 18 years old and able to provide consent

Exclusion criteria:

1. Subjects in whom flexible bronchoscopy is contraindicated
2. Target nodule < 1.0 cm
3. Prior radiation or neo adjuvant chemotherapy of the target nodule/tumor
4. Any comorbidity that the investigator feels would interfere with the safety of the subject or the evaluation of study objectives
5. Pacemaker, implantable cardioverter, or other electronic implantable device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - UT MD Anderson Cancer Center, Houston, Texas
- Toronto General Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RF Ablation
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RF Ablation
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 71 [51 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 5
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: ANET Related Peri-procedural Adverse Events
Description: The incidence of reported adverse events and serious adverse events related to the ANET device or procedure
Time Frame: Day 0
Measure: Number; unit: Adverse Event
Arm/Group | RF Ablation
Number analyzed (Participants) | 6
Adverse Event | 0

ADVERSE EVENTS:
Time Frame: Day 0
Arm/Group | RF Ablation
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Canada (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT03400748/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: United States (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT03400748/Prot_SAP_001.pdf